CLINICAL TRIAL: NCT02101502
Title: Quality Assurance of Obstetrics and Gynecology Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Edessy Mahmoud, Professor, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1781955
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Problems With Access to Health Care
Keywords: Healthcare,educational effectiveness, institutional capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Institutional Capacity (Active Comparator): Questioner for institutional employee about Institutional Capacity
  Interventions: Other: Questioner
- Educational Effectiveness (Active Comparator): Questioner for medical and assistant staffs about Educational Effectiveness
  Interventions: Other: Questioner
- Health-care (Active Comparator): Questioner for medical, assistant staffs and patients about Quality Assurance System in Health-care
  Interventions: Other: Questioner

INTERVENTIONS:
Other: Questioner — Obstetrics and gynecology health problems questionnaire for patients Educational effectiveness special questionnaire for medical staffs Institutional capacity special questionnaire for institution employees

SUMMARY:
This work aimed to prepare the obstetrics and gynecology department for high education and health care accreditation.

DETAILED DESCRIPTION:
For Institutional Capacity and Educational Effectiveness we have used a special questioner for assessment (Met or Not Met Questioner). For Quality Assurance System in Health-care we used a special questioner which contain several items each of them may be A ,B or C. A= structured standards, and are scored as M= Met or N=Not Met or NA=Not Applicable ,The B &C standards are implementation standards . these standards are scored either on the number of observations , documentation of deficiencies , or non compliance with the standards.

ELIGIBILITY:
Inclusion criteria:

* Female patients attending the obstetrics and gynecology department
* Medical and assistant medical staffs
* institutional employees

Exclusion criteria:

* Female patients complaining from disorders not included in the obstetrics and gynecology department activities.
* Male patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quality Assurance | One year and 4 months
  QA=Quality Assurance
  * Institutional Capacity
  * Educational Effectiveness
  * Obstetrical and Gynecological disorders of health care

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Edessy, MD, Principal Investigator — Al-Azhar University; Abd El-Naser Mohammad, MD, Study Chair — Al-Azhar University; Manal Abd El-Aty, MD, Study Chair — Al-Azhar University; Mahmoud Badawi, MSc, Study Chair — Al-Azhar University
Locations (1):
- Al-Azhar University (Assuit), Asyut, Assuit, Egypt